CLINICAL TRIAL: NCT06188793
Title: Evaluation of a Virtual Reality-Directed Brain Gut Behavioral Treatment Inpatient Program for Patients With Inflammatory Bowel Disease
Brief Title: Virtual Reality (VR) -Directed Brain Gut Behavioral Treatment (BGBT) for Inflammatory Bowel Disease (IBD) Inpatients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Shirley Cohen-Mekelburg, Assistant Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00240999
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Virtual reality; Inpatient; Pain; Brain Gut Behavioral Treatment
MeSH Terms: conditions — Inflammatory Bowel Diseases; Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual reality-directed BGBT (Experimental)
  Interventions: Device: Virtual reality-directed BGBT

INTERVENTIONS:
Device: Virtual reality-directed BGBT — Enrolled participants will receive up to 3-days of VR-directed BGBT through several modules including distraction games, mindfulness meditation, breathing exercises, and cognitive behavioral therapy based coaching. Participants will complete questionnaires at various time points and be asked to complete a semi-structured interview post-intervention.

SUMMARY:
The research is studying virtual reality (VR)-directed brain-gut behavioral therapy (BGBT) as a pain treatment option for hospitalized patients with inflammatory bowel disease (IBD). This study is being done to learn if VR-directed BGBT is feasible and acceptable for patients with IBD in addressing pain in the hospital setting.

The study hypothesizes that:

* At least 75% of enrolled participants will complete the VR-directed BGBT inpatient program
* Hospitalized patients with IBD will find VR-directed BGBT acceptable as a pain treatment option in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Inflammatory Bowel Disease and self-reported pain
* Hospitalized for management of IBD (inpatient medicine services at Michigan Medicine)

Exclusion Criteria:

* Patients that do not report pain
* Anticipated length of hospital stay is less than 72 hours
* Patients that have previously had a seizure, loss of awareness, or other symptoms linked to an epileptic condition
* Patients with binocular vision loss
* Patients with an uncontrolled cardiac condition such as an arrhythmia, coronary artery disease, or neurological/cerebrovascular disease.
* Patients that are currently pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the intervention measured as the frequency (percentage) of enrolled participants that complete the VR-directed BGBT inpatient program | 3 days of treatment

SECONDARY OUTCOMES:
Intervention acceptability based on qualitative data and collected from audio-recordings of semi-structured interview | 1 week (semi-structured interview within 1 week of completion of the intervention)
  Patient acceptability will be evaluated through semi-structured interviews within 1 week of completion of the intervention to understand satisfaction, expectations, and experiences with the protocol, including perceived benefits or harms, and barriers to use.
Acceptability using the System Usability Scale - patients | Day 3 (post intervention)
  This is a 10-item question scale that are answered from a range from strongly agree to strongly disagree. Scores range from 0 to 100 with a higher score indicating greater acceptability.
Acceptability using the Treatment Acceptance and Adherence Scale- patients | Day 3 (post intervention)
  This is a 10-item question scale that have a range from disagree strongly- agree strongly.
  Scores range from 10-70 with higher scores indication greater acceptability.

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Cohen-Mekelburg, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gutermuth B, Jordan A, Hodish G, Sturgeon JA, DeJonckheere M, Berinstein JA, Sheehan J, Bishu S, Higgins PD, Cohen-Mekelburg S. Evaluation of a virtual reality-directed brain-gut behavioural treatment inpatient program for patients with inflammatory bowel disease: protocol for a pilot feasibility trial. BMJ Open. 2025 Jul 3;15(7):e098674. doi: 10.1136/bmjopen-2024-098674. PMID 40615149